CLINICAL TRIAL: NCT07007611
Title: The Role of Surgical Resection AND Stereotactic Radiosurgery in PCNS-DLBCL: A Retrospective Analysis of Clinical Benefits
Brief Title: The Role of Surgical Resection AND Stereotactic Radiosurgery in Primary Central Nervous System -Diffuse Large B Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: jiahong Deng (Other)
Responsible Party: Sponsor-Investigator, jiahong Deng, Clinical Professor, Southern Medical University, China
Organization: Southern Medical University, China (Other)
Other Study IDs: NFEC-2025-095
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Primary Central Nervous System Diffusing Large Cell Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- primary central nervous system diffusing large cell lymphoma

SUMMARY:
The objective of this observational study is to understand the long-term impact of surgery and gamma knife treatment on primary central diffuse large B-cell lymphoma. The main questions it aims to answer are:

Can surgery and gamma knife prolong the survival period of patients with primary central diffuse large B-cell lymphoma? Participants who have already incorporated surgery and gamma knife as part of the routine medical care for patients with primary central diffuse large B-cell lymphoma will answer questions about survival period within 5 years.

ELIGIBILITY:
Inclusion Criteria:

pathologically confirmed PCNS-DLBCL complete clinical records detailing treatment methods and surgical approaches.

Exclusion Criteria:

incomplete systemic treatment data loss to follow-up after initial contact prior receipt of whole-brain radiotherapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A retrospective analysis was conducted on data from patients diagnosed with primary central nervous system diffuse large B-cell lymphoma (PCNS-DLBCL) at Nanfang Hospital between December 2006 and December 2023. A total of 76 patients were included in this study, with follow-up continuing until July 2024.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2006-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | December 2006 and December 2023
  The time from diagnosis to death of the patient

IPD SHARING:
Plan to Share IPD: No